CLINICAL TRIAL: NCT04260828
Title: Efficacy and Safety Study of Aspirin for the Prevention of Renal Artery Stenosis in Renal Transplantation Recipients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202102310438
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Renal Transplant
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aspirin (Active Comparator)
  Interventions: Drug: Aspirin 100mg
- Placebo (sugar pill) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aspirin 100mg — Daily active drug administered orally for 3 months.
  Arms: Aspirin
Other: Placebo — Sugar pill administered orally for 3 months.
  Arms: Placebo (sugar pill)

SUMMARY:
The anastomotic and peripheral stenosis of the transplanted kidney artery is one of the most important causes of graft failure in renal transplantation. The injury of vascular intima and the formation of microthrombosis may play a significant role in the stenosis of transplanted renal artery of recipients. Inhibiting this process with aspirin may protects against the stenosis of transplanted renal artery.

This is a prospective, randomized, controlled, clinical trial to investigate the efficacy and safety of prevention of renal artery stenosis in recipients.

ELIGIBILITY:
Inclusion Criteria:

1. The patients with the first renal transplantation were stable;
2. Age ≥ 18 years old;
3. Other anticoagulants and non steroidal anti-inflammatory drugs were not taken at the same time;
4. In the past 3 months, there was no acute cardiovascular and cerebrovascular disease or infection;
5. The rejection of acute and chronic renal transplantation was excluded;
6. The thrombus formation of transplanted kidney was excluded.

Exclusion Criteria:

1. Allergic or intolerable to aspirin;
2. Previous transplant history;
3. Age < 18;
4. Take other anticoagulants or non steroidal anti-inflammatory drugs at the same time;
5. History of active gastrointestinal bleeding or severe peptic ulcer;
6. Patients with bleeding tendency or severe liver disease;
7. Cerebral hemorrhage, cerebral infarction or acute infection occurred within 3 months;
8. Acute and chronic rejection;
9. Thrombus formation of transplanted renal vessels;
10. Any condition that increases the risk of adverse events or discontinuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Renal Artery Stenosis | 2 years
  Renal artery stenosis is defined as the presence of post-transplant renal artery stenosis in recipients evaluated by ultrasonography or renal arteriography.

SECONDARY OUTCOMES:
Renal Allograft Function | 2 years
  Renal allograft function is evaluated by mean estimated glomerular filtration rate(eGFR).
Incidence of Graft Loss | 2 years
  The incidence of kidney failure within 2 years of transplant.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Tian X, Ji B, Niu X, Duan W, Wu X, Cao G, Zhang C, Zhao J, Wang Z, Gu Y, Cao H, Qin T, Shao F, Yan T. Efficacy and safety of low-dose aspirin on preventing transplant renal artery stenosis: a prospective randomized controlled trial. Chin Med J (Engl). 2023 Mar 5;136(5):541-549. doi: 10.1097/CM9.0000000000002574. PMID 36914946